CLINICAL TRIAL: NCT03549663
Title: Random, Open, Control and Monocentric Clinical Research on Tacrolimus Monotherapy for Idiopathic Membranous Nephropathy (IMN)
Brief Title: Tacrolimus Monotherapy for Idiopathic Membranous Nephropathy (IMN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-18-006
Record Dates: First submitted 2018-05-10; First posted 2018-06-08 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Tacrolimus; Prednisone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus monotherapy (Experimental)
  Interventions: Drug: Tacrolimus
- Tacrolimus combined with hormone therapy (Active Comparator)
  Interventions: Drug: Tacrolimus; Drug: Prednisone

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus capsules: 0.5mg/pill, 50 pills/box, AstellasPharma (China) Co., Ltd.; Tacrolimus capsules: 1mg/pill, 50 pills/box, Hangzhou ZhongmeiHuadong Pharmacy Co., Ltd. Start to administer on the randomized grouping day (D0) with an initial dose by weight: initial dose of 0.05-0.075mg/kg/d (bid) following a strict administration interval of 12 hours or fasting or 2 hours after meal. Adjust TAC dose according to 24-hour urine protein, plasma concentration and eGFR changes. It is recommended that plasma trough concentration should be remained at 5-8ng/ml and TAC dose during the whole therapy stage should not be lower than 0.5mg/d. Drugs should be stopped if the 6-month therapy is ineffective. After 6-month therapy, for those whose urine protein achieved complete remission (CR) or partial remission (PR), TAC dose should be reduced gradually with a total therapy duration of 48 weeks.
Drug: Prednisone — Glucocorticoid (prednisone): 5mg/pill, 100 pills/bottle: Shanghai Sine Pharmaceutical Factory Co., Ltd. The initial dose of prednisone should be 0.5mg/kg/d orally (maximum dose of 40mg/d) and administration should be continued for 8-12 weeks; then reduced by the monthly decreased amount of 0.1mg/kg/d till to 0.2mg/kg/d (5-10mg) to maintain. Prednisone should be stopped after administration for the entire 48 weeks.
  Other Names: Glucocorticoid
  Arms: Tacrolimus combined with hormone therapy

SUMMARY:
The trial is a random, open, control and monocentric trial. Mainly to assess the urine protein remission rate of tacrolimus (TAC) monotherapy for idiopathic membranous nephropathy (IMN). Assuming that the urine protein remission rate of 48-week TAC for monotherapy of IMN is not lower than that in treatment group of TAC combined with glucocorticoid, attempt on de-hormonal therapy in the future IMN therapy can be attempted on the basis of the trial results.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 80 years;
2. Those whose clinical manifestation and renal biopsy pathologic diagnosis are IMN (Stages I-IV) with secondary membranous nephropathy excluded;
3. Those who meet any of the following high-risk IMN standards:

   * Urinary protein>8g/24h
   * Serum albumin<25g/l
   * Serum PLA2R levels are 5 times higher than normal
   * eGFR decline rate after confirmed IMN within 6-12 months is ≥30%
   * Patients with serious complications: pulmonary embolism, lower extremity static Vein thrombosis/embolism, acute renal injury, etc.
4. Those without reaching the above high-risk IMN standard, but their course of disease is >6 months without spontaneous remission,and still present nephrotic syndrome;
5. Patients who have signed the informed consent forms.

Exclusion Criteria:

1. Those whose kidney pathological manifestation of interstitial fibrosis is >30%;
2. Those who are positive in active Hepatitis B (including HBsAg, HBeAg and HBcAb or HBsAg, HBeAb and HBC) or serological indexes (HBsAg or/and HBeAg or/and HBcAb) or infected with Hepatitis C, tuberculosis, cytomegalovirus, severe fungal or HIV infection;
3. Those who suffer from untreated active digestive tract ulcer within 3 months before random grouping;
4. Those who suffer from uncured malignant tumor for less than 5 years
5. Those who received glucocorticoid (prednisone or prednisolone), mycophenolatemofetil, tacrolimus, cyclosporine A and other drugs for treatment within 3 months before screen with a course of treatment exceeding 4 weeks or those who received cyclophosphamide (accumulated dose>1.0g);
6. Those whose ALT, AST or total bilirubin content goes beyond 1.5 times above normal upper limit;
7. Those who suffer from combined critical complications such as serious infection or other severe organ disease or dysfunction;
8. Pregnant or lactating women;
9. Those who are known to be allergic to drugs under trial or relevant products;
10. Those who participated in other clinical trials within 3 months before inclusion;
11. The patients who cannot comply with the research proposal as determined by the supervising physician.

Exit criteria

1. Those with incomplete or partial relieved proteinuria for 6 months after treatment;
2. Patients or their legal guardians voluntarily requests to withdraw;
3. Those against the inclusion criteria and exclusion criteria;
4. Those who need to take medications prohibited by the trail;
5. Those with poor compliance or stopping the drug for over 2 weeks;
6. Those with uncontrollable infection;
7. Those whit elevated blood glucose during the treatment, which is still difficult to control after routine treatment by endocrinologists;
8. In the TAC group, the eGFR decreased by >30%, the TAC dose was halved. And the drug concentration and renal function were reviewed after 2 weeks. If the eGFR decreased by <30%, it will continue to be used; if the eGFR still decreased by >30%, the TAC dose continues to halve, or give a minimum dose of 0.5mg / d. And the drug concentration and renal function were reviewed after 2 weeks. If the eGFR decreased by <30%, TAC will continue to be used, otherwise stop the drug;
9. Those whose ALT, AST or bilirubin rises to more than 2 times the upper limit of normal value after treatment, and continues to increase for 2 weeks; those whose ALT, AST or bilirubin rises to more than 2 times the upper limit of normal value after 2 weeks of treatment with liver protection, the drug will be discontinued. If it cannot be recovered after 2 weeks, the patient will withdraw;
10. Those with other unexplained severe comorbidities;
11. Those with pregnancy during treatment;
12. For security reasons, the research sponsor proposed to stop the study;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate of 24-hour urine protein | At week 48
  The proportion of patients with complete remission of 24-hour urine protein in the total evaluated patients. Evaluation criteria of complete remission: post-therapy urine protein level is <0.3g/24h.

SECONDARY OUTCOMES:
Partial remission remission rate of 24-hour urine protein | At week 48
  The proportion of patients with partial remission of 24-hour urine protein in the total evaluated patients. Evaluation criteria of partial remission: post-therapy urine protein decline is >50% compared with the peak value.
PLA2R antibody negative conversion rate | At week 48
  The proportion of patients with PLA2R antibody negative conversion in the total evaluated patients. Evaluation criteria of negative conversion: PLA2R antibody level is <20RU/ml.
Number of patients with adverse events | up to 48 weeks
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Fujun Lin, MD,PhD, Principal Investigator — Shanghai Xinhua Hospital affiliated to Shanghai Jiao Tong University, School of Medicine
Locations (1):
- Shanghai Xinhua Hospital affliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zhu P, Zhou FD, Wang SX, Zhao MH, Wang HY. Increasing frequency of idiopathic membranous nephropathy in primary glomerular disease: a 10-year renal biopsy study from a single Chinese nephrology centre. Nephrology (Carlton). 2015 Aug;20(8):560-6. doi: 10.1111/nep.12542. PMID 26086701
- [Background] Xu X, Wang G, Chen N, Lu T, Nie S, Xu G, Zhang P, Luo Y, Wang Y, Wang X, Schwartz J, Geng J, Hou FF. Long-Term Exposure to Air Pollution and Increased Risk of Membranous Nephropathy in China. J Am Soc Nephrol. 2016 Dec;27(12):3739-3746. doi: 10.1681/ASN.2016010093. Epub 2016 Jun 30. PMID 27365535
- [Background] Hofstra JM, Fervenza FC, Wetzels JF. Treatment of idiopathic membranous nephropathy. Nat Rev Nephrol. 2013 Aug;9(8):443-58. doi: 10.1038/nrneph.2013.125. Epub 2013 Jul 2. PMID 23820815
- [Background] du Buf-Vereijken PW, Branten AJ, Wetzels JF. Idiopathic membranous nephropathy: outline and rationale of a treatment strategy. Am J Kidney Dis. 2005 Dec;46(6):1012-29. doi: 10.1053/j.ajkd.2005.08.020. PMID 16310567
- [Background] KDIGO Clinical Practice Guideline for Glomerulonephritis. Kidney Int 2012, 2: 139-274.
- [Background] Ponticelli C, Zucchelli P, Passerini P, Cesana B, Locatelli F, Pasquali S, Sasdelli M, Redaelli B, Grassi C, Pozzi C, et al. A 10-year follow-up of a randomized study with methylprednisolone and chlorambucil in membranous nephropathy. Kidney Int. 1995 Nov;48(5):1600-4. doi: 10.1038/ki.1995.453. PMID 8544420
- [Background] Ponticelli C, Altieri P, Scolari F, Passerini P, Roccatello D, Cesana B, Melis P, Valzorio B, Sasdelli M, Pasquali S, Pozzi C, Piccoli G, Lupo A, Segagni S, Antonucci F, Dugo M, Minari M, Scalia A, Pedrini L, Pisano G, Grassi C, Farina M, Bellazzi R. A randomized study comparing methylprednisolone plus chlorambucil versus methylprednisolone plus cyclophosphamide in idiopathic membranous nephropathy. J Am Soc Nephrol. 1998 Mar;9(3):444-50. doi: 10.1681/ASN.V93444. PMID 9513907
- [Background] Ramachandran R, Hn HK, Kumar V, Nada R, Yadav AK, Goyal A, Kumar V, Rathi M, Jha V, Gupta KL, Sakhuja V, Kohli HS. Tacrolimus combined with corticosteroids versus Modified Ponticelli regimen in treatment of idiopathic membranous nephropathy: Randomized control trial. Nephrology (Carlton). 2016 Feb;21(2):139-46. doi: 10.1111/nep.12569. PMID 26205759
- [Background] Xu J, Zhang W, Xu Y, Shen P, Ren H, Wang W, Li X, Pan X, Chen N. Tacrolimus combined with corticosteroids in idiopathic membranous nephropathy: a randomized, prospective, controlled trial. Contrib Nephrol. 2013;181:152-62. doi: 10.1159/000348475. Epub 2013 May 8. PMID 23689577
- [Background] Chen M, Li H, Li XY, Lu FM, Ni ZH, Xu FF, Li XW, Chen JH, Wang HY; Chinese Nephropathy Membranous Study Group. Tacrolimus combined with corticosteroids in treatment of nephrotic idiopathic membranous nephropathy: a multicenter randomized controlled trial. Am J Med Sci. 2010 Mar;339(3):233-8. doi: 10.1097/MAJ.0b013e3181ca3a7d. PMID 20220333
- [Background] Zhu LB, Liu LL, Yao L, Wang LN. Efficacy and Safety of Tacrolimus Versus Cyclophosphamide for Primary Membranous Nephropathy: A Meta-Analysis. Drugs. 2017 Feb;77(2):187-199. doi: 10.1007/s40265-016-0683-z. PMID 28084563
- [Background] Praga M, Barrio V, Juarez GF, Luno J; Grupo Espanol de Estudio de la Nefropatia Membranosa. Tacrolimus monotherapy in membranous nephropathy: a randomized controlled trial. Kidney Int. 2007 May;71(9):924-30. doi: 10.1038/sj.ki.5002215. Epub 2007 Mar 21. PMID 17377504
- [Background] Liang Q, Li H, Xie X, Qu F, Li X, Chen J. The efficacy and safety of tacrolimus monotherapy in adult-onset nephrotic syndrome caused by idiopathic membranous nephropathy. Ren Fail. 2017 Nov;39(1):512-518. doi: 10.1080/0886022X.2017.1325371. PMID 28562168
- [Background] Hoxha E, Thiele I, Zahner G, Panzer U, Harendza S, Stahl RA. Phospholipase A2 receptor autoantibodies and clinical outcome in patients with primary membranous nephropathy. J Am Soc Nephrol. 2014 Jun;25(6):1357-66. doi: 10.1681/ASN.2013040430. Epub 2014 Mar 7. PMID 24610926